CLINICAL TRIAL: NCT06087354
Title: Effect of Low Versus Air Oxygen Concentration in In-vitro Maturation With Biphasic Capacitation-IVM (CAPA-IVM) Culture of Human Cumulus-oocyte Complexes in PCOS Patients: a Sibling Oocyte Pilot Study
Brief Title: Low vs. Air Oxygen Concentration CAPA-IVM Culture of Cumulus-oocyte Complexes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/23/DD-BVMD
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-10

CONDITIONS: IVM; PCOS (Polycystic Ovary Syndrome)
Keywords: Low oxygen; CAPA-IVM; Cumulus-oocyte complexes
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Oxygen Concentration CAPA-IVM culture (Experimental): Half of COCs were cultured in the CAPA step and IVM step in a low oxygen concentration (5%) and 6% carbon dioxide at 37 degree
  Interventions: Other: The way of Cumulus-oocyte complexes (COC) CAPA-IVM culture condition
- Air Oxygen Concentration CAPA-IVM culture (Experimental): Half of COCs were cultured in the CAPA step and IVM step in a air oxygen concentration (20%) and 6% carbon dioxide at 37 degree
  Interventions: Other: The way of Cumulus-oocyte complexes (COC) CAPA-IVM culture condition

INTERVENTIONS:
Other: The way of Cumulus-oocyte complexes (COC) CAPA-IVM culture condition — Cumulus-oocyte complexes (COC) will be cultured in CAPA-IVM 24 hrs capacitation followed by 30h maturation. The first group will be cultured in low oxygen concentration (5%Oxygen), 6% carbon dioxide at 37 degree. The second group will be cultured in air oxygen concentration (20%Oxygen), 6% carbon dioxide at 37 degree.

SUMMARY:
IVM with a pre-maturation step, known as capacitation IVM (CAPA-IVM), has demonstrated enhanced maturation of human oocytes in vitro and successful live births. However, CAPA-IVM has shown lower rates of embryo formation when compared to conventional in vitro fertilization/ intra cytoplasmic sperm injection (IVF/ICSI) cycles. To optimize the CAPA-IVM culture system, this pilot study aims to evaluate the impact of low oxygen versus air oxygen concentrations on embryological outcomes in PCOS patients.

DETAILED DESCRIPTION:
Oocyte in vitro maturation (IVM) is an alternative approach to assisted reproductive technology (ART) that has the advantage of minimal stimulation, resulting in reduced hormone-related side effects and risks, especially in women with polycystic ovary syndrome (PCOS). Oocytes retrieved for IVM procedures are derived from a diverse pool of follicles with an average diameter of between 2 and 10mm and are characterized by variable cellular and molecular attributes that indicate their immature status. Therefore, the development of an IVM culture system that could enable and enhance the acquisition and synchronization of meiotic and developmental competence prior to the meiotic resumption is essential for optimizing human IVM protocols.

IVM with a pre-maturation step, known as capacitation IVM (CAPA-IVM), has been shown to improve the competence of human oocytes matured in vitro and result in live births. The pre-maturation culture of CAPA-IVM utilizes C-type natriuretic peptide (CNP), and maturation takes place in the presence of amphiregulin (AREG), both of which are physiological compounds that have been shown to prevent spontaneous meiotic resumption of oocytes (CNP) and enhance oocyte competence (AREG) during IVM.

To date, the results of pilot studies have shown that CAPA-IVM increases the rates of oocyte maturation, good-quality embryos on day 3 and good-quality blastocysts, resulting in a result, a higher embryo yield was obtained compared with standard IVM. Additionally, the reported cumulative live birth rate after use of CAPA-IVM, and its non-inferiority to the cumulative live birth rate with standard in vitro fertilization highlight the clinical utility and potential of this approach. Improvements in the culture system could make CAPA-IVM more effective, but these need to be investigated.

The oxygen concentration during the IVM process plays a crucial role in oocyte maturation. The use of oxygen concentrations higher than physiological levels can lead to cell damage and affect embryo development. Recent studies in mice have suggested using lower oxygen concentrations to improve IVM outcomes. However, the effectiveness of using lower oxygen concentrations in human IVM remains unproven. Therefore, this pilot study aims to compare the effectiveness of lower oxygen concentration conditions versus air oxygen in CAPA-IVM on embryology outcomes in PCOS women.

ELIGIBILITY:
Inclusion Criteria:

* ≤38 years
* Having polycystic ovarian morphology: at least 25 follicles (2-9 mm) throughout the whole ovary and/or increased ovarian volume (>10ml)
* Having at least 20 follicles on the Oocyte Pick-up day
* Patients consent to culture embryos to the blastocyst

Exclusion Criteria:

* Cases with severe male factor (concentration <5 million/ml, cryptozoospermia, azoospermia)
* Oocyte donation
* Pre-implantation genetic testing

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Number of blastocyst | At least 5 days after intra-cytoplasmic sperm injection
  Number of blastocyst obtained

SECONDARY OUTCOMES:
Number of matured oocytes | Two days after oocytes pick-up
  Number of oocytes which have a polar body after maturation
Number of normal fertilized oocytes | 16-18 hours after intra-cytoplasmic sperm injection
  Number of oocytes which have 2 pronuclear
Number of day-3 embryos | At least 3 days after intra-cytoplasmic sperm injection
  Number of day-3 embryos obtained
Number of good-quality day-3 embryos | At least 3 days after intra-cytoplasmic sperm injection
  Number of good quality Day 3 embryos obtained
Number of good-quality blastocyst | At least 5 days after intra-cytoplasmic sperm injection
  Number of good quality blastocyst obtained
Number of vitrified blastocyst | At least 5 days after intra-cytoplasmic sperm injection
  Number of vitrified blastocyst obtained
Positive pregnancy test | At 2 weeks after the completion of the first frozen embryo transfer
  Serum human chorionic gonadotropin level greater than 25 mIU/mL
Clinical pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  At least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Ongoing pregnancy | At 12 weeks' gestation
  Defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after the completion of the first transfer
Implantation rate | 3 weeks after embryo transferred after the completion of the first transfer
  Defined as the number of gestational sacs per number of embryos transferred
Multiple pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Miscarriage | at 12 weeks of gestation after the completion of the first transfer
  pregnancy loss at <12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez F, Le AH, Ho VNA, Romero S, Van Ranst H, De Vos M, Gilchrist RB, Ho TM, Vuong LN, Smitz J. Biphasic in vitro maturation (CAPA-IVM) specifically improves the developmental capacity of oocytes from small antral follicles. J Assist Reprod Genet. 2019 Oct;36(10):2135-2144. doi: 10.1007/s10815-019-01551-5. Epub 2019 Aug 9. PMID 31399916
- [Background] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Smitz J, Gilchrist RB, Norman RJ, Mol BW. In-vitro maturation of oocytes versus conventional IVF in women with infertility and a high antral follicle count: a randomized non-inferiority controlled trial. Hum Reprod. 2020 Nov 1;35(11):2537-2547. doi: 10.1093/humrep/deaa240. PMID 32974672
- [Background] Vuong LN, Le AH, Ho VNA, Pham TD, Sanchez F, Romero S, De Vos M, Ho TM, Gilchrist RB, Smitz J. Live births after oocyte in vitro maturation with a prematuration step in women with polycystic ovary syndrome. J Assist Reprod Genet. 2020 Feb;37(2):347-357. doi: 10.1007/s10815-019-01677-6. Epub 2020 Jan 4. PMID 31902102
- [Background] Preis KA, Seidel GE Jr, Gardner DK. Reduced oxygen concentration improves the developmental competence of mouse oocytes following in vitro maturation. Mol Reprod Dev. 2007 Jul;74(7):893-903. doi: 10.1002/mrd.20655. PMID 17192892
- [Background] Akin N, Ates G, von Mengden L, Herta AC, Meriggioli C, Billooye K, Stocker WA, Ghesquiere B, Harrison CA, Cools W, Klamt F, Massie A, Smitz J, Anckaert E. Effects of lactate, super-GDF9, and low oxygen tension during bi-phasic in vitro maturation on the bioenergetic profiles of mouse cumulus-oocyte complexdagger. Biol Reprod. 2023 Oct 13;109(4):432-449. doi: 10.1093/biolre/ioad085. PMID 37531262